CLINICAL TRIAL: NCT04454086
Title: Healthy New Albany: Breast Cancer Project
Brief Title: Exercise and Diet Counseling Program in Improving Quality of Life in Stage I-III Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Brian Focht, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-17122; NCI-2019-00570 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-07-16; First posted 2020-07-01 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Cancer Survivor; Obesity; Overweight; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: conditions — Obesity; Overweight | interventions — Exercise; Nutrition Assessment; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (exercise program, counseling) (Experimental): Patients undergo aerobic exercise over 10-30 minutes and resistance exercise comprising 1-3 sets of 8-12 repetitions of 10 different exercises over 1 hour for 24 weeks. Patients also receive behavioral activity counseling once a week and nutritional counseling over 30 minutes for 10 sessions after center-based exercise sessions during months 1-2.
  Interventions: Other: Aerobic Exercise; Other: Exercise Counseling; Other: Nutritional Assessment; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Resistance Training

INTERVENTIONS:
Other: Aerobic Exercise — Undergo aerobic exercise
  Other Names: Aerobic Activity
Other: Exercise Counseling — Receive behavioral activity counseling
Other: Nutritional Assessment — Receive nutritional counseling
  Other Names: Dietary Assessment; dietary counseling; nutritional counseling
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Resistance Training — Undergo resistance exercises
  Other Names: Strength Training

SUMMARY:
This trial studies the benefits of an exercise and diet counseling program in improving quality of life in stage I-III breast cancer survivors. Exercise and diet counseling may help improve weight loss and relevant clinical and patient-reported outcomes in overweight or obese breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of delivering a community-based, comprehensive lifestyle weight management (LWM) intervention to 20 overweight or obese breast cancer (BC) survivors.

II. Explore preliminary efficacy of the community-based, comprehensive LWM intervention for producing meaningful improvements in select clinically-relevant anthropometric, fitness, functional, and patient-reported outcomes in BC survivors.

III. Provide the effect size estimates necessary to inform the design of a subsequent R01 application addressing a large scale, optimally powered, randomized controlled, community-based LWM comparative efficacy intervention trial targeting weight loss in BC survivors.

OUTLINE:

Patients undergo aerobic exercise over 10-30 minutes and resistance exercise comprising 1-3 sets of 8-12 repetitions of 10 different exercises over 1 hour for 24 weeks. Patients also receive behavioral activity counseling once a week and nutritional counseling over 30 minutes for 10 sessions after center-based exercise sessions during months 1-2.

After completion of study, patients are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer (stage I-III), within (w/in) 60 months after cessation of active treatment (surgery, chemotherapy, radiation), and may be on continued hormone therapy.
* Overweight/obese (body mass index [BMI] > 25).
* Ability to understand and the willingness to sign a written informed consent.
* Willing and physically able to participate in physical activity.
* Obtain physician consent via primary care physician and/or treating oncologist.

Exclusion Criteria:

* > 60 months post breast cancer therapy.
* Contraindications to exercise.
* Diagnosis of cancer other than breast that is receiving active treatment.
* Currently receiving chemotherapy/radiation.
* Musculoskeletal/neurological disorder inhibiting them from safe exercise.
* Pregnant or nursing women.
* Unable to give informed consent.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Mobility disability | Baseline up to 6 months
  Assessed with the 400-meter walk test. Will be analyzed using paired samples t-tests. Statistical significance will be assumed at p =< 0.05, and results will be based on two-tailed statistical tests. Mean change from baseline, paired sample t-test, and effect size estimates will be calculated for each outcome measure. Analyses will be conducted using the intent-to-treat principle to account for missing data with the last observation carried forward (LOCF) approach, used to impute change across time to be zero. Additionally, effect sizes (Cohen?s d) will be calculated by taking the mean difference and dividing by the pooled standard deviation to determine the magnitude of differences observed for each outcome.

SECONDARY OUTCOMES:
Self-reported physical function | Baseline up to 6 months
  Measure with the abbreviated Late-Life Function and Disability Inventory. Will be analyzed using paired samples t-tests. Statistical significance will be assumed at p =< 0.05, and results will be based on two-tailed statistical tests. Mean change from baseline, paired sample t-test, and effect size estimates will be calculated for each outcome measure. Analyses will be conducted using the intent-to-treat principle to account for missing data with the LOCF approach, used to impute change across time to be zero. Additionally, effect sizes (Cohen?s d) will be calculated by taking the mean difference and dividing by the pooled standard deviation to determine the magnitude of differences observed for each outcome.
Objective functional performance | Baseline up to 6 months
  Using 3 valid and reliable timed performance-related mobility tasks: 400-meter walk (the primary outcome), stair-climb, and lift and carry task. Assessments of Mobility-Related Self-Efficacy to complete each functional task will also be completed with the tests. Will be analyzed using paired samples t-tests. Statistical significance will be assumed at p =< 0.05, and results will be based on two-tailed statistical tests. Mean change from baseline, paired sample t-test, and effect size estimates will be calculated for each outcome measure. Analyses will be conducted using the intent-to-treat principle to account for missing data with the LOCF approach, used to impute change across time to be zero. Additionally, effect sizes (Cohen?s d) will be calculated by taking the mean difference and dividing by the pooled standard deviation to determine the magnitude of differences observed for each outcome.
Balance deficits assessment | Baseline up to 6 months
  Estimate standing and reaching balance using a balance plate. Will be analyzed using paired samples t-tests. Statistical significance will be assumed at p =< 0.05, and results will be based on two-tailed statistical tests. Mean change from baseline, paired sample t-test, and effect size estimates will be calculated for each outcome measure. Analyses will be conducted using the intent-to-treat principle to account for missing data with the LOCF approach, used to impute change across time to be zero. Additionally, effect sizes (Cohen?s d) will be calculated by taking the mean difference and dividing by the pooled standard deviation to determine the magnitude of differences observed for each outcome.
Muscular strength assessement | Baseline up to 6 months
  Using standardized one-repetition maximum testing protocols for the chest press and leg extension exercises. Will be analyzed using paired samples t-tests. Statistical significance will be assumed at p =< 0.05, and results will be based on two-tailed statistical tests. Mean change from baseline, paired sample t-test, and effect size estimates will be calculated for each outcome measure. Analyses will be conducted using the intent-to-treat principle to account for missing data with the LOCF approach, used to impute change across time to be zero. Additionally, effect sizes (Cohen?s d) will be calculated by taking the mean difference and dividing by the pooled standard deviation to determine the magnitude of differences observed for each outcome.
Body composition | Baseline up to 6 months
  Dual-energy x-ray absorptiometry (DEXA) for all outcome measures. The DEXA scans were used to determine total body composition including bone-mineral density, as well as, percentage body fat and fat-free mass for all body regions. Will be analyzed using paired samples t-tests. Statistical significance will be assumed at p =< 0.05, and results will be based on two-tailed statistical tests. Mean change from baseline, paired sample t-test, and effect size estimates will be calculated for each outcome measure. Analyses will be conducted using the intent-to-treat principle to account for missing data with the LOCF approach, used to impute change across time to be zero. Additionally, effect sizes (Cohen?s d) will be calculated by taking the mean difference and dividing by the pooled standard deviation to determine the magnitude of differences observed for each outcome.
Body weight | Baseline up to 6 months
  Measured to the nearest 0.1 kilogram using a calibrated and certified balance beam scale. Will be analyzed using paired samples t-tests. Statistical significance will be assumed at p =< 0.05, and results will be based on two-tailed statistical tests. Mean change from baseline, paired sample t-test, and effect size estimates will be calculated for each outcome measure. Analyses will be conducted using the intent-to-treat principle to account for missing data with the LOCF approach, used to impute change across time to be zero. Additionally, effect sizes (Cohen?s d) will be calculated by taking the mean difference and dividing by the pooled standard deviation to determine the magnitude of differences observed for each outcome.
Quality of life (QOL) surveys using the Rand Short Form Health Survey (SF-12) | Baseline up to 6 months
  The SF-12 questionnaire is a 12 -item scale that assesses the Physical (PCS) and Mental Health (MCS) composite summary scales composed of 6 items each on a 5-point rating scale. PCS and MCS scores range from 0-30 with higher scores indicating more favorable outcomes.
Quality of life (QOL) survey using the Functional Assessment of Cancer Therapy- breast (FACT-B). | Baseline up to 6 months
  The Functional Assessment of Cancer Therapy-Breast is a disease specific measures including the satisfaction with life scale. The Functional Assessment of Cancer Therapy-breast will be used to analyze sample T-tests.
Brief Fatigue Inventory (BFI) | Baseline up to 6 months
  The Brief Fatigue Inventory is a 9-item scale scored on an 11-point rating scale ranging from 0 (no fatigue) to 10 (as bad as you can imagine). Higher scores represent greater levels of fatigue. In this form, there are 5 overarching questions. The first one asks, "Have you felt unusually tired or fatigued in the last week?" which is simply a Yes or No response. The next 4 questions then have answers in terms of a scale. The next 3 have the following sliding scale: 0= No Fatigue, 10= As bad as you can imagine, with 1-9 each representing intermediate responses. For the last question, the scale is: 0= Does not interfere, 10= Completely interferes, with 1-9 representing individual intermediate responses.
Adherence assessment | Up to 6 months
  Will be defined via attendance at prescribed sessions and will be assessed using exercise logs, upon which participants will record all exercise performed at the center or independently. Will be analyzed using paired samples t-tests. Statistical significance will be assumed at p =< 0.05, and results will be based on two-tailed statistical tests. Mean change from baseline, paired sample t-test, and effect size estimates will be calculated for each outcome measure. Analyses will be conducted using the intent-to-treat principle to account for missing data with the LOCF approach, used to impute change across time to be zero. Additionally, effect sizes (Cohen?s d) will be calculated by taking the mean difference and dividing by the pooled standard deviation to determine the magnitude of differences observed for each outcome.
Feasibility measures | Up to 24 weeks
  Descriptive statistics for assessments of recruitment rates, adverse events, and retention rates will be calculated prospectively throughout the trial. Feasibility assessments of participants? satisfaction with the exercise and dietary intervention will also be completed at the end of the 24-week intervention. Will be analyzed using paired samples t-tests. Statistical significance will be assumed at p =< 0.05, and results will be based on two-tailed statistical tests. Mean change from baseline, paired sample t-test, and effect size estimates will be calculated for each outcome measure. Analyses will be conducted using the intent-to-treat principle to account for missing data with the LOCF approach, used to impute change across time to be zero. Additionally, effect sizes (Cohen?s d) will be calculated by taking the mean difference and dividing by the pooled standard deviation to determine the magnitude of differences observed for each outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Focht, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu